CLINICAL TRIAL: NCT03106506
Title: Influence of Connective Tissue Graft Placement on the Volume of Soft Tissue Around Implants Placed in Aesthetic Areas. Randomized Controlled Clinical Trial.
Brief Title: Influence of Connective Tissue Graft Around Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Maria Aparecida Neves Jardini, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: f4vqwv6j
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Recession, Gingival
Keywords: Implants; Conjunctive tissue graft; Prospective study
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: A sample of 40 individuals with esthetic need implants will be used for the study, where the test group (n = 20) will receive tec graft. (N = 20) will receive only the dental implant without the placement of a sub-epithelial-conjunctive tissue graft.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test-implant with graft (Experimental): Patients who received a connective tissue graft around implants
  Interventions: Procedure: Connective tissue graft
- Control-Implant without graft (Active Comparator): Implant installation surgery with cone morse system without the placement of connective tissue graft.
  Interventions: Procedure: Connective tissue graft

INTERVENTIONS:
Procedure: Connective tissue graft — Implant installation surgery with cone morse system with the concomitant placement of autogenous connective tissue.

SUMMARY:
The objective of this randomized controlled clinical study was to evaluate the increase in the volume of peri-implant gingival tissue in implants installed in the aesthetic areas with the use of subepithelial-conjunctive tissue graft, and a sample of 40 individuals with implants Aesthetics where the test group (n = 20) will receive tec graft. (N = 20) will receive only the dental implant without the placement of a tec graft. Epithelial-conjunctival.

DETAILED DESCRIPTION:
Osseointegrated implants have been used since the mid-1950s, and countless studies have ensured the reliability of their use, so the implant has become a common practice among dental surgeons, as the use of implants has increased its complications as well. Accompany the same development, especially when they are installed in aesthetic areas, where deficiency of periimplant gingival tissue is insufficient.

The objective of this randomized controlled clinical study was to evaluate the increase in the volume of periimplant gingival tissue in implants installed in the aesthetic areas with the use of subepithelial conjunctive tissue graft, and a sample of 40 individuals with implants aesthetics where the test group (n = 20) will receive tec graft. (N = 20) will receive only the dental implant without the placement of a tec graft epithelial conjunctival.

In order to analyze the increase of gingival periimplant tissue, pre, trans and postoperative clinical measurements, aesthetic evaluation, patient satisfaction assessment and improvement of the quality of life will be performed and the radiographic measurements will be performed to evaluate the periimplant bone structures and their influence on the results.

These measurements will be performed in the pre-operative (baseline), 6 months postoperatively and 6 months after installation of the definitive crown on the implant, the study will have a power of 80% (p = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 20 years of age systemically healthy , oral hygiene satisfactory,assessed by plaque index Gingival Index and less than 25% (O'Leary et al. 1972).
* Patient requiring one implant in the anterior maxilla (premolar of the premolar).
* Availability of healthy bone tissue or greater than five millimeters, with the view to greater primary stability or equal to 35 Ncm
* agreed to participate in the study and sign a written consent ( Resolution No. 196 of October 1996 and the Code of Professional Ethics Dental - C.F.O. - 179/93)

Exclusion Criteria:

* Smokers;
* Patients with parafunctional habits such as bruxism;
* Pregnant or lactating;
* Patients with systemic diseases uncontrolled (cardiovascular diseases, blood disorders, changes in bone metabolism, immunodeficiencies and diabetes) , contraindicate the surgical procedure.
* Drugs that interfere with wound healing, Drug Related gingival hyperplasia phenytoin (dantalin, dialudon, Epelin, fenital, phenytoin, phenytoin sodium, hidantal), cyclosporine A (Restasis, Sandimmun Neoral Sandimmunmicroral Sigmasporin), blockers of calcium channel, (bezilato of amilodipina hydrochloride, ditiaziem, felodipine, isradipine, lacidipine, lercadinipina hydrochloride, micardipina hydrochloride, nifedipine, risoldipina) Immunosuppressive drugs such as Azathioprine, and Prednisolone, drugs of the class of bisphosphonates(alendronate, zoledronate, ibandronate, risedronate, pamidronate, clodronate, etidronate and clodronate) that reduce the metabolism of osteoclasts , inhibiting bone metabolism;
* Implants in adjacent regions;
* Sites of acute infections;
* Sites with large defects in the buccal bone wall;
* Requiring any sort of bone augmentation procedure;
* Patients in orthodontic treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Gain of peri-implant soft tissue | one year
  It is expected that the association of autogenous connective graft to the placement of cone-morse platform implants in aesthetic areas allows a greater gain of peri-implant soft tissue and better aesthetic results after the installation of definitive prostheses than in the other proposed groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jardini, Doctor, Study Director — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- São Jose Dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No